CLINICAL TRIAL: NCT05172752
Title: A University-Community Partnership to Reduce Exposure to Disinfection Byproducts In Appalachia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Hoover (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Anna Hoover, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 62921; 1R01ES032396-01 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-12-29 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Disinfection By-products
Keywords: Community-engaged; Appalachia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citizen Science Training (Other): Study participants in this condition will participate in training and in-home sampling for disinfection by-products.
  Interventions: Other: Citizen Scientist Training Program
- Stakeholder Consultation Core Membership (Other): Study participants in this condition will participate in quarterly meetings and deliberative activities of the project's Stakeholder Consultation Core.
  Interventions: Other: Stakeholder Consultation Core Program

INTERVENTIONS:
Other: Citizen Scientist Training Program — Citizen Scientist Training Program Participants is a three year training and in-home sampling program for disinfection byproducts. Participants will be trained and assessed based on their experience in the training program.
  Arms: Citizen Science Training
Other: Stakeholder Consultation Core Program — Stakeholder Consultation Core Program Participants is a five year assessments where participants will participate in quarterly meetings and deliberative activities related to disinfection byproducts. Participants will be assessed based on their experience in the program.
  Arms: Stakeholder Consultation Core Membership

SUMMARY:
Appalachian Kentuckians in Martin and Letcher Counties are grappling with a health-threatening drinking water crisis arising from exposures to disinfection by-products (DBPs). DBPs include trihalomethanes (THMs), haloacetic acids (HAAs), chlorate, and other compounds that have been associated with a variety of adverse health effects, including increased risk of bladder cancer and cardiovascular birth defects. This study implements a multi-stakeholder, multi-method approach to improve understanding of, characterize spatial and temporal variations in, and reduce exposure to DBPs in these Appalachian Kentucky counties.

ELIGIBILITY:
Inclusion Criteria:

* Located in Martin or Letcher County water districts
* At least 18 years old
* Able to read/speak in English

Exclusion Criteria:

* Located outside of Martin or Letcher County water districts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Environmental Health Literacy (EHL) - Knowledge | Baseline, 5-years
  Study participants will complete pre-/post-surveys of disinfection byproducts-related knowledge. Participants will answer 21 questions with multiple choice or fill in the blank response options that will be assessed for correctness/completeness.
Change in Environmental Health Literacy (EHL) - Attitudes/Behaviors | Baseline, 5-years
  Study participants will complete pre-/post-surveys of disinfection byproducts-related attitudes. Participants will answer 9 questions related attitudes/behaviors with a five-point Likert scale, ranging from Strongly Disagree to Strongly Agree, where Strongly Agree indicates a greater likelihood for the behavior/more positive attitude.
Change in participant network density | Baseline, 5-years
  The proportion of direct ties within the network as compared to the number of possible ties as measured by an unbounded social media analysis.
Change in participant centrality | Baseline, 5-years
  The influence of each individual within the network (i.e., betweenness and degree centrality) as measured by an unbounded social media analysis.
Change in participant reciprocity | Baseline, 5-years
  The number of reciprocal ties, which is the extent to which individuals within the network recognize each other as valued resources/collaborators as measured by an unbounded social media analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Hoover, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No